CLINICAL TRIAL: NCT00452309
Title: Validation of a Correction Factor for Measurement of an Accurate Ankle-Brachial Index in the Seated Position
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Summit Doppler Systems, Inc. (Industry)
Other Study IDs: IRB 06-1007
Record Dates: First submitted 2007-03-25; First posted 2007-03-27 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; pad; ankle brachial index; abi
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to test a correction factor which would allow ankle brachial indexes taken in the seated position to accurately predict an ankle brachial index taken in the supine position.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a highly prevalent medical condition. Patients with PAD are usually diagnosed on the basis of a simple diagnostic procedure know as the ankle-brachial index (ABI). The ABI is the ratio of ankle pressure to arm pressure after measurement of blood pressures in the arms and legs using a hand-held Doppler device. In order for the ABI measurement to be accurate, the test is conducted with the patient in the supine position. This eliminates the influence of hydrostatic pressure on the ankle and toes which can lead to a falsely elevated reading. Unfortunately, many patients are unable to lie supine for ABI measurement, including: the wheel-chair bound, patients with degenerative disease of the spine or arthritis with chronic back pain, and patients with advanced cardiopulmonary disease and orthopnea.

Given the importance of detecting PAD across a broad spectrum of patients, there is a need to identify a mechanism for reliable measurement of the ABI for patients who cannot lie supine. The purpose of this study is to test a correction factor for the effects of hydrostatic pressure on the lower extremities to allow for accurate ABI calculation in the seated position.

100 Subjects with suspected arterial disease in the vascular lab will be enrolled. Arm, ankle, and toe pressure measurements will be made in the supine and seated positions. The seated ankle pressures will be corrected for hydrostatic pressure using a mechanical formula. The ABI and toe brachial index (TBI) will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 60 years of age
* Ambulatory outpatient
* Referred to non-invasive Vascular Laboratory for evaluation of suspected arterial disease.

Exclusion Criteria:

* Unable to give informed consent
* Unable to lie supine for at least 15 minutes

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather L Gornik, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Gornik HL, Garcia B, Wolski K, Jones DC, Macdonald KA, Fronek A. Validation of a method for determination of the ankle-brachial index in the seated position. J Vasc Surg. 2008 Nov;48(5):1204-10. doi: 10.1016/j.jvs.2008.06.052. Epub 2008 Sep 30. PMID 18829231